CLINICAL TRIAL: NCT04902027
Title: A Multicenter, Open-label, Single-arm, Phase Ib Study to Evaluate Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Recurrent/Metastatic Head and Neck Cancers
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Recurrent/Metastatic Head and Neck Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-016
Record Dates: First submitted 2021-03-18; First posted 2021-05-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Head and Neck Cancer; Metastatic Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Subjects with Rrecurrent/metastatic Head and Neck Cancers will receive 20 mg/m2 Mitoxantrone Hydrochloride Liposome every 21 days (a cycle) for a maximum of 8 cycles
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV)

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV) — All subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2, IV, on day 1 of each 21-day cycle (q3w).

SUMMARY:
This is a multicenter, open-label, single-arm, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with recurrent/metastatic Head and Neck Cancers

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with recurrent/metastatic head and neck cancers. At least 30 subjects will be recruited in this study. The subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2 by an intravenous infusion (IV), every 21 days (q3w, 1 cycle). All patients will receive the treatment until disease progression, intolerable toxic reaction, death, or withdrawa by investigator or patient decision (a maximum of 8 cycles). Delays in drug administration is allowed from the cycle 2, however, the delays should be no more than 3 weeks. Dose adjustments after the cycle 2 is permitted, and the minimum dose is 12mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. . Age ≥18, female or male;
3. Histologically confirmed diagnosis of head and neck squamous cell carcinoma (including nasopharyngeal carcinoma)
4. Fail to respond to or progressed on at least one line of the standard therapy;
5. At least one measurable lesion according to RECIST v1.1;
6. ECOG performance status of 0 to 1;
7. AEs from the previous treatment have resolved to ≤ Grade 1 based on

Exclusion Criteria:

1. History of allergy to mitoxantrone hydrochloride or any excipients of the study drug;
2. Untreated or symptomatic central nervous system (CNS) metastases;
3. History of allotransplantation;
4. Life expectancy < 3 months
5. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or other active viral infection;
6. Serious infection or interstitial pneumonia within 1 week prior to the first dose administration;
7. Use of other anticancer treatment within 4 weeks prior to the first dose administration;
8. Enrolled in any other clinical trials within 4 weeks prior to the first dose administration;
9. Major surgery within 3 months prior to the first dose administration, or have a surgical schedule during the study period;
10. Thrombosis or thromboembolism within 6 months prior to screening;
11. History of, or known additional malignant tumor within 3 years, except for tumors have been cured and have not recurred, and carcinoma in situ;
12. Impaired cardiac function or serious cardiac disease
13. Previous treatment with adriamycin or other anthracyclines, and the total cumulative dose of prior adriamycin or equivalent is >350 mg/m2
14. Pregnant or lactating female;
15. Serious and/or uncontrolled systemic diseases;
16. Not suitable for this study as decided by the investigator due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
adverse events (AEs),,graded according to the NCI CTCAE version 5.0 | from the initiation of the first dose to 28 days after the last dose
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
(best total response) (BOR) | From the enrollment to the final documentation of response of the last subject ( at least 6 weeks between follow-up and enrolment
  To investigate the preliminary antitumor efficacy
duration of response (DoR) | From the enrollment to CR, PR, PD, death, lost to follow-up, withdrawal, or study end, assessed up to 2 years
  To investigate the preliminary antitumor efficacy
progression-free survival (PFS) | from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 2 years
  To investigate the preliminary antitumor efficacy
overall survival (OS) | from date of enrollment until date of first death from any cause, assessed up to 2 years
  To investigate the preliminary antitumor efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, MD, Study Chair — Cancer Prevention Center, Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China